CLINICAL TRIAL: NCT07269834
Title: Effects of a Workplace Exercise Program on Stress, Burnout, and Quality of Life in Radiologic Technologists
Brief Title: Workplace Exercise and Well-Being in Radiologic Technologists
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pedro Ramalho (Other)
Collaborators: University of Beira Interior (Other)
Responsible Party: Sponsor-Investigator, Pedro Ramalho, Principal Investigator, University of Beira Interior
Organization: University of Beira Interior (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EXER-RAD-2025
Record Dates: First submitted 2025-11-25; First posted 2025-12-08 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Occupational Stress or Workplace Stress; Burnout; Quality of Life; Exercise Training; Radiologists; Health Promotion
MeSH Terms: conditions — Occupational Stress; Burnout, Psychological

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group (Experimental): Participants are involved in a workplace exercise program.
  Interventions: Behavioral: Workplace Exercise Program
- Control group (Other): Non-exercise group
  Interventions: Other: Control (Non-exercise)

INTERVENTIONS:
Behavioral: Workplace Exercise Program — Participants complete a six-week workplace exercise program comprising structured sessions based on methodologies described in previous studies (Alqhtani et al., 2023; Gelfman et al., 2024). Sessions are conducted three times per week, twice per day, with each session lasting approximately 15 to 20 minutes.
  The program includes exercises primarily performed in a standing position and aims to improve flexibility, balance, and strength.
  Flexibility training: Static and dynamic stretching exercises performed three times per week, 1-2 sets per exercise, held for 10-15 seconds each.
  Balance training: Static and dynamic balance exercises performed three times per week, 1-3 sets per exercise, for 10-20 repetitions or 10-20 seconds over a 3-6 meter distance.
  Strength training: Bodyweight and resistance exercises using auxiliary equipment (e.g., elastic bands), performed three times per week, 1-3 sets per exercise, 8-15 repetitions per set, with a slow to moderate tempo.
  Arms: Exercise group
Other: Control (Non-exercise) — Participants in the control (non-exercise) group maintain their usual work routines and will not participate in any structured exercise sessions during the study period.
  Arms: Control group

SUMMARY:
Radiologic technologists often face demanding work conditions that contribute to elevated stress levels and increased burnout risk, ultimately affecting both their well-being and professional effectiveness. Workplace exercise initiatives have shown potential benefits for improving physical and psychological health; however, experimental research targeting this specific occupational group is still scarce. The main aim of this study is to evaluate the effects of a structured workplace exercise intervention on perceived stress, burnout, and quality of life among radiologic technologists. The secondary objective is to assess the effects of a detraining period on the same outcomes following completion of the exercise program.

ELIGIBILITY:
Inclusion Criteria:

* Healthy radiographers (diagnostic and therapeutic imaging technologists)
* Currently employed in the radiology department of the participating hospital
* Voluntary participation with signed informed consent

Exclusion Criteria:

* Presence of major musculoskeletal, cardiovascular, or neurological conditions that contraindicate physical exercise;
* Pregnancy;
* Unavailability to attend regular exercise sessions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2025-08-14 (Actual); Primary Completion 2025-10-30 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Changes in Quality of Life Levels | From baseline to 6 weeks (end of the exercise program)
  The World Health Organization Quality of Life - BREF (WHOQOL-BREF) was used. The Portuguese version was adapted and validated by Canavarro et al. (2007).
Changes in Burnout Levels | From baseline to 6 weeks (end of the exercise program)
  The Copenhagen Burnout Inventory (CBI), developed by Kristensen et al. (2005) and adapted for the Portuguese population by Fonte (2011), was used to assess burnout levels.
Changes in Perceived Stress Levels | From baseline to 6 weeks (end of the exercise program)
  The Perceived Stress Scale (PSS) was developed by Cohen, Kamarck, and Mermelstein (1983) and aims to measure an individual's subjective perception of stress intensity in their life - specifically, the degree to which situations are evaluated as unpredictable, uncontrollable, or overwhelming. The Portuguese version of the PSS-10 was validated by Trigo et al. (2010).

SECONDARY OUTCOMES:
Changes in quality of life, stress, and burnout | End of intervention (week 6) and after 4 weeks of detraining (week 10)
  WHOQOL-BREF; Perceived Stress Scale; Copenhagen Burnout Inventory (CBI)

CONTACTS AND LOCATIONS:
Locations (1):
- Local Health Unit of Castelo Branco (ULSCB), Castelo Branco, Portugal

IPD SHARING:
Plan to Share IPD: Undecided
De-identified data that support the findings of this study may be made available from the corresponding author upon reasonable request and following approval by the Ethics Committee.